CLINICAL TRIAL: NCT01710540
Title: AN OPEN LABEL, BALANCED, RANDOMIZED, TWO-TREATMENT, TWO-PERIOD, TWO-SEQUENCE, CROSSOVER, SINGLE ORAL DOSE, BIOEQUIVALENCE STUDY OF METFORMIN GSK 850 MG TABLETS MANUFACTURED BY SAVIPHARM J.S.C, VIETNAM AND GLUCOPHAGE® 850 MG TABLETS MANUFACTURED BY MERCK SANTE S.A.S.2, RUE DU PRESSOIR VERT-45400 SEMOY-FRANCE AND BE REGISTERED IN VIETNAM IN HEALTHY, ADULT, HUMAN MALE SUBJECTS UNDER FASTING CONDITION
Brief Title: BE Study of Metformin GSK 850mg
Acronym: BA/BE 198/11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 116728
Record Dates: First submitted 2012-09-27; First posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin GSK 850mg (Other): open label, crossover, two period, two treatment, two sequence, single dose of Metformin 850mg
  Interventions: Other: Metformin GSK 850mg; Other: Gluocophage 850mg
- Glucophage 850mg (Other): open label, crossover, two period, two treatment, two sequence, single dose
  Interventions: Other: Metformin GSK 850mg; Other: Gluocophage 850mg

INTERVENTIONS:
Other: Metformin GSK 850mg — EVALUATE BIOEQUIVALENCE BETWEEN METFORMIN 850 MG TABLETS MANUFACTURED BY SAVIPHARM J.S.C, VIETNAM AND GLUCOPHAGE® 850 MG TABLETS MANUFACTURED BY MERCK SANTE S.A.S.2, RUE DU PRESSOIR VERT-45400 SEMOY-FRANCE AND BE REGISTERED IN VIETNAM IN HEALTHY, ADULT, HUMAN MALE SUBJECTS UNDER FASTING CONDITION
Other: Gluocophage 850mg — EVALUATE BIOEQUIVALENCE BETWEEN METFORMIN 850 MG TABLETS MANUFACTURED BY SAVIPHARM J.S.C, VIETNAM AND GLUCOPHAGE® 850 MG TABLETS MANUFACTURED BY MERCK SANTE S.A.S.2, RUE DU PRESSOIR VERT-45400 SEMOY-FRANCE AND BE REGISTERED IN VIETNAM IN HEALTHY, ADULT, HUMAN MALE SUBJECTS UNDER FASTING CONDITION

SUMMARY:
A randomized, balanced, open label, crossover, two period, two treatment, two sequence, single dose, oral bioequivalence study under fasting condition. It is a pivotal study to demonstrate the bioequivalence of Metformin 850 mg tablets manufactured by Savipharm J.S.C, Vietnam and Glucophage® 850 mg tablets of Merck Sante, France, in healthy adult human male subjects under fasting condition.

DETAILED DESCRIPTION:
Sample Size Estimation Assuming the formulation ratio (T/R) 95-105% and with the maximum observable intra subject variability for Metformin is 22% (based on literature), a sample size of 29 subjects would be sufficient to prove bioequivalence between the two formulations with power of at least 90%. Hence, total 32 subjects will be enrolled in the study considering withdrawal and dropouts.

Screening procedures: Demographic data, medical and medication histories, complete physical examination, height, weight and BMI as well as 12 lead ECG, chest X-ray [PA view], vital signs [blood pressure, pulse rate, respiratory rate and oral temperature], hematology, biochemistry, HIV 1 & 2, Hepatitis B and C, RPR test for Syphilis and urine analysis will be done at screening.

Urine drug screen, Liver chemistry test and breath alcohol test to be done prior to each check-in.

Breath alcohol test to be done prior to each ambulatory visit blood collection. Liver chemistry test to be done at the end of each period. Housing: The study subjects will be housed at least 11 h prior to drug administration until after the 24 h blood sampling in each study period. The housing will be followed by one ambulatory visits [36.0 hr post dose] for each period.

Washout: At least 7 days, but not exceeding 14 days between two dosing days. Treatment arms: Test: A single dose of Metformin 500 mg tablet manufactured by Savipharm J.S.C, Vietnam.

Reference: A single dose of Glucophage® 500 mg tablet of Merck Sante, France Drug administration: As per the randomization schedule, one tablet of either test or reference product will be orally administered to each subject in each period in sitting posture, after an overnight fast of at least 10 h.

To avoid hypoglycemic episodes, the investigational products will be administered with 240 mL of a 20% glucose solution in water, followed by 60 mL of the glucose solution administered every 15 min for up to 4 h after dosing.

Subjects will be instructed not to chew or crush the tablet but should be swallowed. Compliance for dosing will be assessed by identification of subjects with subject ID card, identification of label on investigational product to confirm correct allocation of treatment and checking the oral cavity immediately after dosing.

Restrictions: Subjects will remain in upright position [sitting or ambulatory] for two hours after dosing in each period except when clinically indicated to change the posture. The subjects will fast for at least 10 h prior to dosing and 4 h post-dose. Water will be permitted ad libitum except for 1 h before and until 1 h after post dose. During 1 hr post dose water restriction a, 60 mL of 20% glucose solution will be administered every 15 min to the study subjects.

In each period of the study, 18 blood samples of 6 mL each will be collected in K2EDTA vacutainers via an indwelling catheter placed in one of the forearm veins. Heparin-lock technique will be used to prevent clotting of blood in the indwelling catheter. Before each in-house blood sample is drawn through catheter, 0.5 mL of blood will be discarded so as to purge the heparin containing blood sample in the catheter. Blood can also be collected by direct venipuncture in case of cannula blockage, during ambulatory visits or for any other practical reasons. The two pre-dose blood samples will be collected within a period of 1 h before the drug administration. The post-dose blood samples will be collected at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 36.0 h. The 36.0 h post dose blood samples will be collected during ambulatory visits by direct venipuncture. Immediately after collection of blood, the sample will be kept in ice bath. After collecting the blood samples from all the subjects at each sampling time point, samples will be centrifuged at 4oC with 3500 rpm for 10 minutes. The plasma samples will be separated and stored in pre-labeled polypropylene tubes at -70 ± 10°C pending assay. The time interval between sample collection and the start of centrifugation should not exceed more than 45 minutes. The blood sample collection, processing and analysis will be done under sodium monochromatic light.

The total volume of blood drawn including the volume necessary for the laboratory tests, PK sample analysis and the volume of blood discarded before each in house blood draw will be about 250 mL per subject for the entire study.

Subjects monitoring: Brief physical examination and vital signs [blood pressure, pulse rate and oral temperature] will be carried out and recorded at each check-in and at check-out. Vital signs [blood pressure and pulse rate] will also be recorded before dosing of investigational products, between 2 - 3, 9 - 10 and 36.0 h post dose. Vital signs should be done in sitting position after rest of at least 5 minutes. Physical examination and measurement of vital signs can also be carried out at any time during the conduct of the study if the Investigator/Doctor feels it necessary. In case of abnormality in pre-dose vital signs, Investigator based on his medical judgement will take the decision whether to dose the subject or not. During vitals recording each subject will be asked about his well-being. Also subject well-being questionnaire will be performed at 1.0 and 5.0 h post dose.

Post-study Procedures: Safety evaluation [complete physical examination, vital signs, hematology [except blood grouping & Rh typing] and biochemistry] will be done at the end of the clinical part of the study. In case of any withdrawals during the study safety assessment will be done at the time of withdrawal. In case of dropouts subjects will be asked to visit the facility to undergo safety assessments.

Pharmacokinetic Parameters: Cmax, Tmax, AUC0-t, AUC0-∞, AUC%_Extrap, Kel and t1/2 Analytical Methods: Metformin in plasma will be estimated using validated LC-MS/MS method.

Statistical Methods: Statistical analyses will be done using SAS® version 9.2 or higher. Analysis of variance [ANOVA] for log-transformed pharmacokinetic parameters [Cmax, AUC0-t and AUC0-∞], two one-sided tests [Schuirmann] for bioequivalence, power, ratio and 90% confidence interval for log-transformed pharmacokinetic parameters - Cmax, AUC0-t and AUC0-∞ will be performed.

Standards for Bioequivalence: The calculated 90% Confidence Interval for the test to reference ratio of Metformin should fall within the range of 80%-125% for log transformed Cmax, AUC0-t and AUC0-∞ for the conclusion of bioequivalence.

Adverse Events The investigator or site staff is responsible for detecting, documenting and reporting events that meet the definition of an AE or SAE.

AEs will be collected from the start of Study Treatment and until the follow-up contact. Medical occurrences that begin prior to the start of study treatment but after obtaining informed consent may be recorded on the Medical History/Current Medical Conditions CRF.

SAEs will be collected over the same time period as stated above for AEs. However, any SAEs assessed as related to study participation (e.g. study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication will be recorded from the time a subject consents to participate in the study up to and including any follow-up contact. All SAEs will be recorded and reported to the sponsor within 24 hours.

Investigators are not obligated to actively seek AEs or SAEs in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he considers the event reasonably related to the study treatment or study participation, the investigator would promptly notify the sponsor.

All serious adverse events will be informed to the sponsor within 24 hrs and to the IEC within 7 working days. Any unexpected serious adverse event (SAE) occurring during a clinical trial should be communicated promptly (within 14 calendar days) by the Sponsor/CRO to the Licensing Authority.

Any follow-up information on a previously reported SAE will also be reported to the sponsor within 24 hours.

If the investigator does not have all information regarding an SAE, he/she will not wait to receive additional information before notifying the sponsor of the event and completing the appropriate data collection tool. The investigator will always provide an assessment of causality at the time of the initial report.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male human subjects within the age range of 18 to 45 years inclusive.
* Weight not less than 50 kg.
* Normal BMI [18.5 to 24.99 kg/m2 inclusive].
* Willingness and capability to provide written informed consent to participate in the study.
* Free of significant diseases or clinically significant abnormal findings based on medical history, physical examination, laboratory evaluations, 12-lead ECG, Chest X-ray [PA view].
* Absence of disease markers of HIV 1 and 2, Hepatitis B and C and Syphilis.
* AST, ALT, alkaline phosphatase and bilirubin </=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* ECG normal for morphology and measurements. QTcB or QTcF < 450 msec or QTc < 480 msec in subjects with Bundle Branch Block, based on an average from three ECGs obtained over a brief recording period.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed below. This criterion must be followed from the time of the first dose of study medication until one week of last dose administration.

  * Condom plus partner use of a highly effective contraceptive such as occlusive cap (diaphragm or cervical/vault cap) plus spermicidal agent (foam/gel/film/cream/suppository), oral contraceptive, injectable progesterone, implant of etonogestrel or levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, or intrauterine device.

OR

* Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* History or presence of significant: Cardiovascular, pulmonary, hepatic, renal, hematological, gastro-intestinal, endocrine, immunologic, dermatologic, neurological, psychiatric disease.
* History or presence of significant:

  * Alcohol dependence, alcohol abuse during past one year.
  * Drug abuse [Marijuana [THC], Cocaine, Morphine, Benzodiazepines, Barbiturates and Amphetamine] for the last 6 months.
  * Smoking of more than 5 cigarettes per day or consumption of other forms of tobacco containing products.
  * Asthma, urticaria or other allergic type reactions after taking aspirin or any other drug.
  * Ulceration or history of gastric and / or duodenal ulcer.
  * Jaundice in the past 6 months.
* Bleeding disorder.
* Allergy to the test drug or any drug chemically similar to the drug or to the excipients of the products under investigation.
* Donation of 500 mL or more blood within 8 weeks prior to receiving the first dose of study drug.
* Subjects who have participated in another clinical study in the past 3 months prior to commencement of this study.
* Any difficulty in accessibility of forearm veins for cannulation or blood sampling.
* Refusal to abstain from food for at least 10 h prior to drug administration and for at least 4 h post dose in each period.
* Refusal to abstain from fluid for at least 1 h prior to and 1 h post each dose except 20 % glucose solution given after dosing.
* Positive breath alcohol test result found on the day of check-in.
* Positive urine test result for drug of abuse found on the day of check-in.
* History of difficulty in swallowing tablet.
* Use of any concomitant medication [including over-the-counter products, vitamins etc.] for 14 days preceding the study drug administration.
* Use of drugs which induce or inhibit metabolizing enzymes within 30 days prior to receiving the first dose of study medication.

Other Eligibility Criteria Considerations To assess any potential impact on subject eligibility with regard to safety, the investigator must refer to the product data sheet for detailed information regarding warnings, precautions, contraindications, adverse events, and other significant data pertaining to the product being used in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, AUC0-t, AUC0-∞, AUC%_Extrap, Kel and t1/2 | 7days
  Statistical analyses will be done using SAS® version 9.2 or higher. Analysis of variance [ANOVA] for log-transformed pharmacokinetic parameters [Cmax, AUC0-t and AUC0-∞] and two one-sided tests [Schuirmann] for bioequivalence will be performed. Power, ratio and 90% confidence interval for log-transformed pharmacokinetic parameters - Cmax, AUC0-t and AUC0-∞ will be calculated. The calculated 90% Confidence Interval for the test to reference ratio of Metformin should fall within the range of 80%-125% for log transformed Cmax, AUC0-t and AUC0-∞ for the conclusion of bioequivalence.

SECONDARY OUTCOMES:
Safety profile | 14 days
  The Principal Investigator will monitor safety data throughout the course of the study. A qualified medical doctor experienced in conducting bioequivalence study will be available during housing in the clinical center. Subjects will be monitored throughout the study period for occurrence of any adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline